CLINICAL TRIAL: NCT01207973
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamic of Multiple Rising Oral Doses (50, 100, 200 and 350 mg qd and 100 mg Bid for 12 Days) of BI 113823 as Tablet in Male and Female Patients With Osteoarthritis of the Knee (Randomised, Double-blind, Placebo-controlled Within the Dose Groups, Clinical Phase I)
Brief Title: Safety, Tolerability, Pharmacokinetics and -Dynamics of Multiple Rising Oral Doses of BI 113823 in Patients Patients With Osteoarthritis of the Knee
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1272.2; 2010-018541-62 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-09-22; First posted 2010-09-23 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-11

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

ARMS (1):
- BI 113823 (Experimental): 5 dose-groups of multiple oral doses of BI 113823
  Interventions: Drug: BI 113823

INTERVENTIONS:
Drug: BI 113823 — 5 dose-groups of multiple oral doses of BI 113823

SUMMARY:
The objective of the study is to investigate the safety and tolerability of BI 113823 in male and female patients with osteoarthritis, following oral administration of BI 113823 with repeated rising doses.

ELIGIBILITY:
Inclusion criteria patients with osteoarthritis

Exclusion criteria

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2010-09; Primary Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Safety (Physical examination) | 15 days
Safety (Vital signs) | 15 days
Safety (12-lead ECG) | 15 days
Safety (Clinical laboratory tests) | 15 days
Safety (Adverse Events) | 15 days
Tolerability (Assessment of tolerability by investigator) | 15 days

SECONDARY OUTCOMES:
Measures of pharmacodynamic effects | 15 days
Standard pharmacokinetic parameters for single dose and steady state conditions will be assessed | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1272.2.1 Boehringer Ingelheim Investigational Site, München, Germany